CLINICAL TRIAL: NCT05121181
Title: Reaching Consensus on the Definition of Difficult Cholecystectomy Among Spanish Experts. A Delphi Project. Qualitative Study
Brief Title: Reaching Consensus on the Definition of Difficult Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Candido Fernando Alcazar-Lopez (Other)
Collaborators: Hospital Universitario Getafe (Other); Complejo Hospitalario Universitario de Badajoz (Other); Hospital Miguel Servet (Other)
Responsible Party: Sponsor-Investigator, Candido Fernando Alcazar-Lopez, Doctor, Hospital General Universitario de Alicante
Organization: Hospital General Universitario de Alicante (Other)
Other Study IDs: 0
Record Dates: First submitted 2021-07-22; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: delphi project — delphy study

SUMMARY:
Being able to predict the difficulty of a preoperatively can increase safety and improve results. However, a consensus must be reached regarding the definition of a cholecystectomy as "difficult". The aim of this study is to achieve a national expert consensus.

Methods A Delphi study was conducted. Based on the literature, a history of biliary pathology, preoperative clinical, analytical, and radiological data, and intraoperative findings were selected and rated on a Likert scale.

Inter-rater agreement was defined as "unanimous" when 100% of the participants gave an item the same the Likert scale rating; as "consensus" when ≥80% agreed; as "majority" when the agreement was ≥70%.

DETAILED DESCRIPTION:
A Delphi study was conducted. Inter-rater agreement was defined as "unanimous" when 100% of the participants gave an item the same the Likert scale rating; as "consensus" when ≥80% agreed; as "majority" when the agreement was ≥70%.

ELIGIBILITY:
Inclusion Criteria:

* Spanish surgeons
* experts in laparoscopic cholecystectomy, with more than 10 years of experience

Exclusion Criteria:

* not Spanish
* not experts in laparoscopic cholecystectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spanish experts in laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
consensus | 1 month
  Likert scale: 1: "totally disagree", 2: "disagree", 3: "neither agree nor disagree", 4: "agree", and 5: "totally agree".

CONTACTS AND LOCATIONS:
Overall Officials: Alba Manuel Vázquez, Dr, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Alba Manuel Vázquez, Madrid, Spain